CLINICAL TRIAL: NCT06333860
Title: A Phase 4 Multicenter, Randomized, Open-label, Efficacy Assessor Blinded Study of Risankizumab Compared to Deucravacitinib for the Treatment of Adult Subjects With Moderate Plaque Psoriasis Who Are Candidates for Systemic Therapy
Brief Title: A Study to Learn How Safe and Effective Risankizumab is When Compared to Deucravacitinib to Treat Participants With Moderate Plaque Psoriasis and Who Need to Try Systemic Treatment (Works Throughout the Whole Body)
Acronym: IMMpactful
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M24-541
Record Dates: First submitted 2024-03-21; First posted 2024-03-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Moderate Plaque Psoriasis
Keywords: risankizumab; deucravacitinib
MeSH Terms: interventions — risankizumab; deucravacitinib

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Period A: Arm 1 Risankizumab Dose A (Experimental): Participants will be centrally randomized at the Baseline (Day 1) visit to receive Risankizumab as a single SC injection
  Interventions: Drug: Risankizumab
- Period A: Arm 2 Deucravacitinib Dose A (Experimental): Participants will be centrally randomized at the Baseline (Day 1) visit to receive Deucravacitinib orally once per day until the day prior to Week 16
  Interventions: Drug: Deucravacitinib
- Period B: Arm 2a Risankizumab Dose A (Continued) (Experimental): Participants initially randomized to risankizumab (Arm 1) will continue to receive risankizumab as a single SC injection at Weeks 16, 28, and 40
  Interventions: Drug: Risankizumab
- Period B: Arm 2b Deucravacitinib Dose A (Experimental): Participants initially randomized to Deucravacitinib (Arm 2) will be re-randomized at the Week 16 visit to receive Deucravacitinib orally once per day up to Week 52
  Interventions: Drug: Deucravacitinib
- Period B: Arm 2a Risankizumab Dose A (Experimental): Participants initially randomized to Deucravacitinib (Arm 2) will be re-randomized at the Week 16 visit to receive Risankizumab as a single SC injection at Weeks 16, 20, 32, and 44
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Solution for Subcutaneous (SC) injection
  Arms: Period A: Arm 1 Risankizumab Dose A; Period B: Arm 2a Risankizumab Dose A; Period B: Arm 2a Risankizumab Dose A (Continued)
Drug: Deucravacitinib — Oral tablet
  Arms: Period A: Arm 2 Deucravacitinib Dose A; Period B: Arm 2b Deucravacitinib Dose A

SUMMARY:
Psoriasis is a long-term skin disease which causes red, itchy, scaly patches most commonly on the knees, elbows, scalp, and torso (chest, back, and abdomen). In participants with psoriasis, certain skin cells multiply much faster and the skin can develop rough patches that may be red or white with scales. There are many types of psoriasis, but plaque psoriasis is the most common. The exact cause of psoriasis is unknown, but researchers think it may be caused by the body's immune system not working properly.

This study is designed to enroll 336 participants 18 years of age and older with have been diagnosed with moderate chronic plaque psoriasis for at least 6 months prior to Baseline (Day 1) and who have not previously been treated with a biologic treatment (natural substance that is made by using living cells in a laboratory). This is a Phase 4, randomized, open-label, assessor blinded, active comparator study with 2 Parts. Phase 4 studies test treatments that have already been approved to treat patients with a condition or disease. This study is open-label, which means that both participants and study doctors know which study treatment is given to participants

Participants will be administered subcutaneous (SC) treatment of risankizumab every 12 weeks for up to 44 weeks or provided deucravacitinib oral tablets to be taken once daily.

There may be higher treatment burden for participants in this trial compared to their standard of care (due to study procedures). Participants will attend regular (weekly, monthly) visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participant with a diagnosis of chronic plaque psoriasis (PsO) with or without psoriatic arthritis, for at least 6 months prior to Baseline.
* Stable moderate chronic plaque psoriasis at both Screening and Baseline as defined as:

  * Body Surface Area (BSA) ≥ 10% and ≤ 15%,
  * Psoriasis Area and Severity Index (PASI) ≥ 12, and
  * Static Physician Global Assessment (sPGA) = 3 (moderate) based on a 5-point scale (0 to 4).
* Participant must be a candidate for systemic therapy as assessed by the investigator
* Psoriasis inadequately controlled by topicals, phototherapy and/or systemic treatments (including, but not limited to, methotrexate, apremilast, cyclosporine A, corticosteroids, and/or cyclophosphamide)

Exclusion Criteria:

* Participants with any form of PsO other than chronic plaque PsO (e.g., pustular PsO, palmoplantar pustulosis, acrodermatitis of Hallopeau, erythrodermic, or guttate PsO).
* Participants with a history of current drug-induced PsO or a drug-induced exacerbation of preexisting PsO.
* Participants with a history of active ongoing inflammatory skin diseases other than PsO (with or without PsA) that could interfere with the assessment of PsO (e.g., hyperkeratotic eczema).
* Participants with a history of severe renal insufficiency defined as creatinine clearance < 30 mL/min and/or requiring hemodialysis or peritoneal dialysis.
* Participantswith a history of clinically significant (per investigator's judgment) drug or alcohol abuse within the last 6 months.
* Participants with a history of an allergic reaction or significant sensitivity to constituents of the study drugs (and its excipients) and/or other products in the same class.
* Participants who have had major surgery performed within 12 weeks prior to randomization or planned during the conduct of the study (e.g., hip replacement, aneurysm removal, stomach ligation).
* Participants with evidence of:

Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, defined as:

* HBV: Hepatitis B surface antigen (HBs Ag) positive (+) test or detected sensitivity on the HBV DNA PCR qualitative test for subjects who are hepatitis B core antibody (HBc Ab) positive (+) (and for hepatitis B surface antibody [HBs Ab] positive [+] participants where mandated by local requirements).
* HCV: HCV RNA detectable in any participant with anti-HCV antibody (HCV Ab).
* Human immunodeficiency virus (HIV), defined as confirmed positive anti-HIV Ab test and considered to have unstable disease (Unless meeting criteria for stable disease) Participants with HIV with no history of AIDS-defining conditions AND stable disease for at least 6 months prior to screening can be enrolled. Criteria for stable disease is achieved if all below criteria are met. Documentation of "stable disease" can be done at the Screening visit or by documentation of labs performed within 1 month of the Randomization visit, in addition to the subject's medical history.
* On stable antiretroviral therapy;
* Viral load (HIV RNA) below the lower limit of quantification by a validated and approved plasma HIV-1 RNA quantitative assay;
* CD4+ T cell count ≥ 500 cells/μL.

  - Participants with any of the following medical diseases or disorders:
* Recent (within past 6 months) cerebrovascular accident or myocardial infarction;
* History of an organ transplant which requires continued immunosuppression;
* Active or suspected malignancy or history of any malignancy within the last 5 years except for successfully treated non-melanoma skin cancer (NMSC) or localized carcinoma in situ of the cervix.
* Prior history of suicide attempt at any time in the subject's lifetime prior to signing the informed consent and randomization, or major depression or suicidal ideation or attempt requiring hospitalization within the last 3 years prior to signing the informed consent.
* Hereditary problems of galactose intolerance, total lactase deficiency, or glucose-galactose malabsorption.

  - Participants who received within 30 days prior to Baseline any:
* Other systemic immunomodulating treatments (including, but not limited to:

  e.g., methotrexate, apremilast, cyclosporine A, corticosteroids, cyclophosphamide, tofacitinib [Xeljanz®]);
* Other systemic PsO treatments (e.g., retinoids, fumarates, any other drug known to possibly benefit PsO);
* Photochemotherapy (e.g., PUVA), phototherapy (e.g., UVB) or prolonged exposure or use of tanning booths or ultraviolet light sources.

  * Participants who received within 14 days prior to Baseline any topical treatment for PsO or any other skin condition (including, but not limited to: e.g., corticosteroids, vitamin D analogues, vitamin A analogues, pimecrolimus, retinoids, salicyl vaseline, salicylic acid, lactic acid, tacrolimus, tar, urea, or anthralin).
  * Participants who have been treated with any strong cytochrome P450 enzyme inducers (e.g., rifampin, phenobarbital, carbamazepine, phenytoin, St. John's Wort) within 30 days or 5 half-lives of start of treatment with deucravacitinib.
  * Participants who received any live viral or bacterial vaccine within 4 weeks prior to the first dose of study drug, or expect the need for live vaccination during study participation including at least 147 days (21 weeks or as guided by the local risankizumab label [if approved], whichever is longer) after the last dose of risankizumab or at least 30 days after the last dose of deucravacitinib.
  * Participants who have been treated with any investigational drug within 30 days or 5 half-lives of the drug (whichever is longer) prior to the first dose of study drug or be currently enrolled in another interventional clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Period A: Percentage of Participants Achieving 90% Improvement in Psoriasis Area Severity Index (PASI) Score (PASI 90) | At Week 16
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Period A: Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) Score of 0 (Clear) or 1 (Almost Clear) with at least 2-grade improvement from Baseline | Baseline, Week 16
  The static Physicians Global Assessment (sPGA) is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA composite score ranges from 0 to 4 and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5.
Period B: Percentage of Participants Achieving 90% Improvement in Psoriasis Area Severity Index (PASI) Score (PASI 90) in the Intent to Treat Population for non-responders in Period B (ITT_B_NR). | At Week 52
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 90 is defined as at least a 90% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Number of Participants Experiencing Adverse Events (AEs) | Baseline up to 73 Weeks
  An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not the event is considered causally related to the use of the product.

SECONDARY OUTCOMES:
Period A: Percentage of Participants Achieving 100% Improvement in Psoriasis Area Severity Index (PASI) Score (PASI 100) | At Week 16
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 100 is defined as at least a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Period A: Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) Score of 0 with at least 2-grade improvement from Baseline | Baseline. Week 16
  The static Physicians Global Assessment (sPGA) is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA composite score ranges from 0 to 4 and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5.
Period B: Percentage of Participants Achieving 100% Improvement in Psoriasis Area Severity Index (PASI) Score (PASI 100) among participants in the ITT_B_NR Population | At Week 52
  The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis. PASI 100 is defined as at least a 100% reduction in PASI score compared with the Baseline PASI score. The percent reduction in score is calculated as (PASI score at Baseline - score at follow-up visit) / PASI score at Baseline * 100.
Period B: Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) Score of 0 with at least 2-grade improvement from Baselineamong participants in the ITT_B_NR Population. | At Week 52
  The static Physicians Global Assessment (sPGA) is an assessment by the investigator of the overall disease severity at the time of evaluation. Erythema (E), induration (I), and desquamation (D) are scored on a 5-point scale ranging from 0 (none) to 4 (severe). The sPGA composite score ranges from 0 to 4 and is calculated as Clear (0) = 0 for all three; Almost clear (1) = mean >0, <1.5; Mild (2) = mean ≥1.5, <2.5; Moderate (3) = mean ≥2.5, <3.5; and Severe (4) = mean ≥3.5.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (88):
- United States (39):
  - Total Skin and Beauty Dermatology Center /ID# 263011, Birmingham, Alabama
  - Advanced Research Associates - Glendale /ID# 263621, Glendale, Arizona
  - Clear Dermatology & Aesthetics Center /ID# 263626, Scottsdale, Arizona
  - Dermatology Trial Associates /ID# 264480, Bryant, Arkansas
  - First OC Dermatology /ID# 263003, Fountain Valley, California
  - Integrative Skin Science and Research /ID# 264504, Sacramento, California
  - Physioseq, LLC /ID# 265035, Sacramento, California
  - Medderm Associates Dermatology /ID# 263858, San Diego, California
  - Southern California Dermatology /ID# 263021, Santa Ana, California
  - Clearlyderm Dermatology - West Boca /ID# 264963, Boca Raton, Florida
  - Driven Research /ID# 263002, Coral Gables, Florida
  - Skin Care Research - Hollywood /ID# 263877, Hollywood, Florida
  - International Dermatology Research /ID# 264911, Miami, Florida
  - Lenus Research and Medical Group /ID# 263886, Miami, Florida
  - Wellness Clinical Research - Miami Lakes /ID# 263887, Miami Lakes, Florida
  - Skin Care Research - Tampa /ID# 263880, Tampa, Florida
  - Advanced Clinical Research Institute /ID# 263878, Tampa, Florida
  - University Dermatology and Vein Clinic, LLC /ID# 263028, Chicago, Illinois
  - Arlington Dermatology /ID# 263001, Rolling Meadows, Illinois
  - Dawes Fretzin, LLC /ID# 264578, Indianapolis, Indiana
  - MetroBoston Clinical Partners /ID# 263860, Boston, Massachusetts
  - University of Michigan Health System - Ann Arbor /ID# 265233, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan - Clinton Township Office /ID# 264968, Clinton Township, Michigan
  - Dermatology and Skin Center of Lees Summit /ID# 263560, Lee's Summit, Missouri
  - Physician Research Collaboration, LLC /ID# 263568, Lincoln, Nebraska
  - Skin Cancer and Dermatology Institute - Reno /ID# 263697, Reno, Nevada
  - StracSkin, PLLC /ID# 263024, Portsmouth, New Hampshire
  - Oregon Dermatology & Research Center /ID# 263674, Portland, Oregon
  - Clinical Partners /ID# 263862, Johnston, Rhode Island
  - Health Concepts /ID# 263016, Rapid City, South Dakota
  - Arlington Research Center, Inc /ID# 263908, Arlington, Texas
  - Bellaire Dermatology Associates /ID# 263897, Bellaire, Texas
  - U.S. Dermatology Partners - Cedar Park /ID# 263906, Cedar Park, Texas
  - Dermatology Treatment and Research Center /ID# 267071, Dallas, Texas
  - Texas Dermatology Research Center /ID# 264487, Plano, Texas
  - Dermatology Clinical Research Center of San Antonio /ID# 263869, San Antonio, Texas
  - Center for Clinical Studies - Clear Lake /ID# 263009, Webster, Texas
  - Center for Clinical Studies - Clear Lake /ID# 263917, Webster, Texas
  - Premier Clinical Research /ID# 263679, Spokane, Washington
- Australia (6):
  - Paratus Clinical Research Woden /ID# 263120, Phillip, Australian Capital Territory
  - Premier Dermatology /ID# 263119, Kogarah, New South Wales
  - The Skin Hospital - Sydney /ID# 263634, Sydney, New South Wales
  - Veracity Clinical Research /ID# 263091, Woolloongabba, Queensland
  - Skin Health Institute /ID# 263116, Carlton, Victoria
  - Sinclair Dermatology - Melbourne /ID# 262997, East Melbourne, Victoria
- Belgium (3):
  - Cliniques Universitaires UCL Saint-Luc /ID# 263106, Brussels, Brussels Capital
  - UZ Gent /ID# 263107, Ghent, Oost-Vlaanderen
  - CHU de Liege /ID# 263108, Liège
- Canada (6):
  - Dermatology Research Institute - Blackfoot Trail /ID# 264476, Calgary, Alberta
  - Beacon Dermatology Inc /ID# 264266, Calgary, Alberta
  - Wiseman Dermatology Research /ID# 265317, Winnipeg, Manitoba
  - Toronto Dermatology Centre /ID# 264273, Toronto, Ontario
  - Private Practice - Dr. Kim Papp Clinical Research /ID# 264269, Waterloo, Ontario
  - Private Practice - Dr. Angelique Gagne-Henley /ID# 264267, Saint-Jérôme, Quebec
- Germany (7):
  - Universitaetsklinikum Freiburg /ID# 263069, Freiburg im Breisgau, Baden-Wurttemberg
  - Hautarztpraxis Langenau /ID# 263070, Langenau, Baden-Wurttemberg
  - Beldio Research GmbH /ID# 263073, Memmingen, Bavaria
  - Dermatologie Mahlow /ID# 263072, Blankenfelde-Mahlow, Brandenburg
  - Fachklinik Bad Bentheim /ID# 263066, Bad Bentheim, Lower Saxony
  - Universitaetsklinikum Muenster /ID# 263061, Münster, North Rhine-Westphalia
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 263955, Berlin
- Greece (5):
  - University General Hospital Attikon /ID# 263421, Athens, Attica
  - General Hospital Andreas Syggros /ID# 263418, Athens, Attica
  - General Hospital Andreas Syggros /ID# 263708, Athens, Attica
  - Hospital of Skin and Venereal Diseases- Thessaloniki /ID# 263419, Thessaloniki
  - Papageorgiou General Hospital /ID# 263414, Thessaloniki
- Hungary (5):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 263484, Debrecen, Hajdú-Bihar
  - Derm-surg /ID# 263799, Kaposvár, Somogy County
  - Semmelweis Egyetem /ID# 263483, Budapest
  - UNO Medical Trials /ID# 263478, Budapest
  - Szegedi Tudomanyegyetem /ID# 263800, Szeged
- Italy (4):
  - IRCCS Istituto Clinico Humanitas /ID# 263466, Rozzano, Lombardy
  - Duplicate_Azienda Ospedaliera Universitaria Federico II /ID# 264034, Naples, Napoli
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 263986, Bologna
  - Azienda Ospedaliero Universitaria Pisana /ID# 263468, Pisa
- Netherlands (2):
  - Amsterdam UMC, locatie AMC /ID# 263550, Amsterdam, North Holland
  - Spaarne Gasthuis - Hoofddorp /ID# 263165, Hoofddorp, North Holland
- Puerto Rico (5):
  - Private Practice - Dr. Alma Cruz /ID# 263212, Carolina
  - Pan American Center for Oncology Trials /ID# 263206, Rio Piedras
  - Clinical Research Puerto Rico /ID# 263213, San Juan
  - GCM Medical Group, PSC /ID# 263198, San Juan
  - Mindful Medical Research /ID# 263201, San Juan
- Spain (3):
  - Hospital General Universitario de Alicante Doctor Balmis /ID# 262977, Alicante
  - Hospital Clinic de Barcelona /ID# 263040, Barcelona
  - Hospital Universitario de La Princesa /ID# 262980, Madrid
- United Kingdom (3):
  - Victoria Hospital /ID# 262984, Kirkcaldy, Fife
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 262981, London, Greater London
  - Northern Care Alliance NHS Group /ID# 262983, Salford

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M24-541